CLINICAL TRIAL: NCT06072703
Title: A Randomized, Sham-Controlled Clinical Trial Evaluating Individualized Neuromodulation of Cortical Regions Involved in Neurogenic Overactive Bladder in Multiple Sclerosis
Brief Title: Neuromodulating Cortical Regions Involved in Neurogenic Bladder in MS
Acronym: MSBLADDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rose Khavari, M.D., MD/PI, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00035884
Record Dates: First submitted 2023-05-11; First posted 2023-10-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Neurogenic Bladder; Multiple Sclerosis; Overactive Bladder
Keywords: Neurogenic bladder; Functional Neuroimaging; repetitive Transcranial Magnetic Stimulation (rTMS); Neuromodulation
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Multiple Sclerosis; Urinary Bladder, Overactive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Intervention Model: 2:1 active: sham assignment, with an optional OLE phase
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking: Double (participants and principal investigator and co-investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): 1 Hz (LF) and 10 Hz (HF) rTMS stimulation will be delivered at 90% of the resting motor threshold for 40 min each week day for two weeks.
  Interventions: Device: Magstim Rapid2 System
- Sham rTMS (Sham Comparator): Low-frequency (1Hz) active rTMS stimulation will be delivered with an inert "sham" stimulation coil for 40 min each week day for two weeks.
  Interventions: Device: Magstim Rapid2 System

INTERVENTIONS:
Device: Magstim Rapid2 System — The Magstim Rapid2 system is the most commonly used magnetic stimulation system for rTMS clinical studies and therapeutic investigations, capable of selectively inducing, modulating or suppressing neuronal activity. This rTMS device will be used along with the D70 Alpha Coil package, which includes an active coil ideal for focal rTMS and a sham coil, The placebo coil looks identical to its active version and replicates pulse noise without producing the magnetic field necessary to modulate cortical neurons. Additionally, the investigators will be utilizing the StimGuide navigation system (currently available at the HMRI) to accurately target the proposed regions of interest.
  The Magstim Rapid2 system is indicated to be used in Multiple Sclerosis patients as target users with lower urinary tract symptoms such as urinary frequency, urinary urgency, urinary incontinence and voiding dysfunction.
  Other Names: Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Neurogenic overactive bladder (NOAB), characterized by urinary frequency, urgency or urgency incontinence symptoms occurring during the storage phase of the bladder, is the most common urinary complaint in multiple sclerosis (MS). Current management options for NOAB in MS have limited efficacy and considerable adverse effects, which underscores the significance of this study and highlights the need for better, less invasive therapies. This novel study investigates brain therapeutic targets that could shift the focus of NOAB management in MS from a bladder-centric focus to brain restoration; specifically modulating the brain regions identified in the prior functional magnetic resonance imagining studies. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive brain stimulation that can modulate neurons (excite or inhibit) to improve the connectivity of the regions of interest (ROI). The preliminary data demonstrate, for the first time, significant improvement in bladder symptoms in ten women with MS who have voiding dysfunction following multifocal transcranial magnetic stimulation without any treatment-related adverse effects.

This randomized double-blind, sham-controlled single center clinical trial with an optional open-label extension (OLE) phase is designed to evaluate the effects of targeted rTMS in women with MS and NOAB by investigating restorative reorganization of brain function The main purpose of this study is to determine the effects of individualized repetitive Transcranial Magnetic Stimulation (rTMS) for improving overactive bladder symptoms such as urinary frequency and urgency with or without incontinence in individuals with multiple sclerosis (MS). Patients will undergo initial screening that includes a demographics information, physical exam, past medical and surgical history, medication list, urine pregnancy test (female subjects with childbearing potential), and completion of questionnaires to confirm the eligibility of patients. All eligible patients will be required to complete a functional MRI scan followed by locating the regions of interest through neural navigation system and finally receiving 10 treatment sessions.

Since this is a randomized trial, some patients will receive active treatment/ therapy sessions while others will only receive sham or placebo treatments. The total duration to complete all treatment sessions and follow up visits is approximately 4-5 months.

DETAILED DESCRIPTION:
Neurogenic overactive bladder (NOAB), characterized by urinary frequency, urgency or urgency incontinence symptoms occurring during the storage phase of the bladder, is the most common urinary complaint in multiple sclerosis (MS). Current management options for NOAB in MS have limited efficacy and considerable adverse effects, which underscores the significance of this study and highlights the need for better, less invasive therapies. This novel study investigates brain therapeutic targets that could shift the focus of NOAB management in MS from a bladder-centric focus to brain restoration; specifically modulating the brain regions identified in the prior functional magnetic resonance imagining studies. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive brain stimulation that can modulate neurons (excite or inhibit) to improve the connectivity of the regions of interest (ROI). The preliminary data demonstrate, for the first time, significant improvement in bladder symptoms in ten women with MS who have voiding dysfunction following multifocal transcranial magnetic stimulation without any treatment-related adverse effects.

This randomized double-blind, sham-controlled single center clinical trial with an optional open-label extension (OLE) phase is designed to evaluate the effects of targeted rTMS in women with MS and NOAB by investigating restorative reorganization of brain function and improvement of urinary frequency, urgency and incontinence.

Investigators hypothesize that cortical alterations in bladder volume sensing and their response to stimulation contribute to NOAB symptoms in MS, and that improving the response to bladder distention (ROI within circuits 1 and 2) with neuronavigated rTMS can restore brain activity and improve symptoms (frequency, urgency, and incontinence). Investigators will test this hypothesis with the following specific aims:

Aim 1: To determine the clinical effects of neuronavigated and multifocal active/sham rTMS in women with MS and NOAB Aim 2: To assess the neuroimaging restorative effects of neuronavigated active/sham rTMS in women with MS and NOAB Aim 3: To assess the long-term safety and therapeutic effects of repeated rTMS in women with MS and NOAB who participate in the OLE phase (which subjects from both groups will be invited to enter at the 3-month follow up).

Efforts to improve the current knowledge of brain contribution to lower urinary tract function and the development of an individualized, noninvasive, and effective treatment modality at the level of the brain will greatly impact the quality of life for individuals with MS and subsequently others with OAB, whether neurogenic or non-neurogenic

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age)
* Clinically stable MS defined as ExpandedDisability Status Score (EDSS) ≤ 7.5without exacerbation worsening in the preceding 6 months prior to study entry
* Neurogenic Lower Urinary Tract Dysfunction symptoms ≥ 3 months with NBSS total ≥ 15
* Individuals with Montreal Cognitive Assessment (MoCA) score >10 will be eligible
* At least one bladder storage symptoms (e.g., urinary frequency, urinary urgency, nocturia with or without incontinence) indicated by OAB -AT≥ 8
* Individuals with active urinary tract infection (UTI) will be treated and will be enrolled after negative urinalysis

Exclusion Criteria:

* Pregnant/planning to become pregnant or nursing
* Urodynamic findings of bladder outlet obstruction
* Baclofen or other intrathecal pumps, Pacemakers.
* History of seizure disorder (SZ), immediate family of SZ disorder, in addition to individuals who are taking any medications such as (bupropion) Wellbutrin or substances (ex: heavy alcohol use) that would lower seizure threshold will be excluded.
* History of bipolar disorder, or individuals who are taking medications that can exacerbate the condition such as tricyclic antidepressants, selective serotonin reuptake inhibitors, serotonin-nor-epinephrine reuptake inhibitors, anti-psychotics, lithium, bupropion (Wellbutrin) and antihistamines will be excluded.
* All intracranial lesions and hemorrhagic stroke will be excluded
* History of moderate to severe heart disease or unstable angina
* History of Autonomic Dysreflexia
* History of interstitial cystitis, pelvic radiation
* Intra-detrusor botulinumtoxinA (BTX-A) injection over the past 6 months
* Incarcerated patients will be excluded.
* Active sacral nerve stimulation (SNS) device or any other spinal stimulators
* Indwelling urethral or suprapubic catheter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in subjective clinical outcomes following treatment - Neurogenic Bladder Symptom Score (NBSS) Questionnaire | Baseline, 1 week after, 1 month after and 3 months after rTMS treatment
  The subjective clinical assessment includes changes in validated questionnaires. This assessment has 24 questions that measure bladder symptoms across 3 different domains: incontinence (score range: 0-29), storage and voiding (score range: 0-22), and consequences (score range: 0-23); the highest score is associated with worse symptoms. The last question focuses on quality of life scored from 0 (pleased) to 4 (unhappy). The investigators report raw scores here for all domains and QoL.
Changes on patient reported outcomes following treatment - 2 day bladder diary | Baseline, 1 week after, 1 month after and 3 months after rTMS treatment
  Here the investigators evaluate changes on the number of times that symptoms associated with neurogenic overactive bladder occur in a 24hr period after rTMS treatment. Reported outcomes by patients include the number of times the following occur: voids, nocturia, severe urgency episodes, and urgency urinary incontinence episodes.

SECONDARY OUTCOMES:
Changes in brain activation patterns following rTMS treatment - functional MRI imaging | Baseline and 1 week after rTMS treatment
  Effect of rTMS treatment in increasing/decreasing activation in ROIs known to be involved in bladder function measured by changes in blood-oxygen-level-dependent (BOLD) signal.
Changes in objective clinical outcomes following treatment - Bladder Capacity | Baseline, 1 week after, 1 month after and 3 months after rTMS treatment
  The objective clinical assessment includes changes in bladder capacity (mL), which is assessed by collecting both post void residual (PVR) and voided volume (both in mL) in participants after treatment as compared to baseline.
Changes in %Post-Void Residual/Bladder Capacity (PVR/BC) following treatment | Baseline, 1 week after, 1 month after and 3 months after rTMS treatment
  Percentage of PVR in proportion to the bladder capacity will be measured before the intervention and post intervention at 1 and 3 months follow up and will be compared between active and sham neurostimulation groups

OTHER OUTCOMES:
Changes in subjective clinical outcomes following treatment - American Urological Association Symptom Score (AUASS) Questionnaire | Baseline, 1 week after, 1 month after and 3 months after rTMS treatment
  The subjective clinical assessment includes changes in validated questionnaires. This assessment has 8 questions and is used to assess how bothersome urinary symptoms are and quality of life. The investigators report raw scores here for questions pertaining to voiding symptoms. Questions 1-7 have the following score range: 0-5 (with the highest score associated with worse symptoms). The last question pertains to quality of life and has a score range of: 0-6 (with the highest score associated with very reduced quality of life).
Changes in subjective clinical outcomes following treatment - Incontinence Impact Questionnaire Short Form (IIQ-7) | Baseline, 1 week after, 1 month after and 3 months after rTMS treatment
  The subjective clinical assessment includes changes in validated questionnaires. This assessment has 7 questions and is used to assess the impact urine leakage has on a patient's activities, relationships, and feelings. Each question has the following score range: 0-3 (with the highest score associated with higher symptom distress).
Changes in subjective clinical outcomes following treatment - Overactive Bladder (OAB) Awareness Tool | Baseline, 1 week after, 1 month after and 3 months after rTMS treatment
  The subjective clinical assessment includes changes in validated questionnaires. The OAB Awareness Tool assessment has 9 questions. It allows participants to score symptoms and illustrates how these symptoms may be affecting quality of life. Questions 1-8 have a score range of 0-5 (the higher the score the more bothersome the symptom is) and the last questions asks if the participant is male (if so 2 points are added to the total score).

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Khavari R, Elias SN, Boone T, Karmonik C. Similarity of functional connectivity patterns in patients with multiple sclerosis who void spontaneously versus patients with voiding dysfunction. Neurourol Urodyn. 2019 Jan;38(1):239-247. doi: 10.1002/nau.23837. Epub 2018 Oct 12. PMID 30311665
- [Background] Khavari R, Elias SN, Pande R, Wu KM, Boone TB, Karmonik C. Higher Neural Correlates in Patients with Multiple Sclerosis and Neurogenic Overactive Bladder Following Treatment with Intradetrusor Injection of OnabotulinumtoxinA. J Urol. 2019 Jan;201(1):135-140. doi: 10.1016/j.juro.2018.07.066. PMID 30076906
- [Background] Khavari R, Tran K, Helekar SA, Shi Z, Karmonik C, Rajab H, John B, Jalali A, Boone T. Noninvasive, Individualized Cortical Modulation Using Transcranial Rotating Permanent Magnet Stimulator for Voiding Dysfunction in Women with Multiple Sclerosis: A Pilot Trial. J Urol. 2022 Mar;207(3):657-668. doi: 10.1097/JU.0000000000002297. Epub 2021 Oct 25. PMID 34694911
- [Background] Khavari R, Karmonik C, Shy M, Fletcher S, Boone T. Functional Magnetic Resonance Imaging with Concurrent Urodynamic Testing Identifies Brain Structures Involved in Micturition Cycle in Patients with Multiple Sclerosis. J Urol. 2017 Feb;197(2):438-444. doi: 10.1016/j.juro.2016.09.077. Epub 2016 Sep 21. PMID 27664581
- [Background] Shi Z, Tran K, Karmonik C, Boone T, Khavari R. High spatial correlation in brain connectivity between micturition and resting states within bladder-related networks using 7 T MRI in multiple sclerosis women with voiding dysfunction. World J Urol. 2021 Sep;39(9):3525-3531. doi: 10.1007/s00345-021-03599-4. Epub 2021 Jan 29. PMID 33512570
- [Background] Tran K, Karmonik C, Boone TB, Khavari R. Are White Matter Tract Integrities Different in Multiple Sclerosis Women With Voiding Dysfunction? Female Pelvic Med Reconstr Surg. 2021 Jan 1;27(1):e101-e105. doi: 10.1097/SPV.0000000000000830. PMID 32265400
- [Background] Tran K, Shi Z, Karmonik C, John B, Rajab H, Helekar SA, Boone T, Khavari R. Therapeutic effects of non-invasive, individualized, transcranial neuromodulation treatment for voiding dysfunction in multiple sclerosis patients: study protocol for a pilot clinical trial. Pilot Feasibility Stud. 2021 Mar 24;7(1):83. doi: 10.1186/s40814-021-00825-z. PMID 33757581
- [Derived] Salazar BH, Hoffman KA, Lincoln JA, Karmonik C, Rajab H, Helekar SA, Khavari R. Evaluating noninvasive brain stimulation to treat overactive bladder in individuals with multiple sclerosis: a randomized controlled trial protocol. BMC Urol. 2024 Jan 25;24(1):20. doi: 10.1186/s12894-023-01358-8. PMID 38273296